CLINICAL TRIAL: NCT03597828
Title: The Effect on Respiratory Function of Monitored Anesthesia Care With Dexmedetomidine in Patients Undergoing Diagnostic or Therapeutic Pleuroscopy
Brief Title: Respiratory Function of Dexmedetomidine in Patients Undergoing Pleuroscopy
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Sidiropoulou, Assistant Professor of Anesthesiology, Attikon Hospital
Other Study IDs: DEXPLEURO
Record Dates: First submitted 2018-06-27; First posted 2018-07-24 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Pleural Effusions, Chronic; Pleural Effusion, Malignant; Pleural Diseases
Keywords: Monitored Anesthesia Care; Pleuroscopy; dexmedetomidine; fentanyl; midazolam; sedation
MeSH Terms: conditions — Pleural Effusion; Bronchiolitis Obliterans Syndrome; Pleural Effusion, Malignant; Pleural Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DEXMEDETOMIDINE: Dexmedetomidine infusion for pleuroscopy sedation. Rescue drugs will be midazolam for inadequate sedation and fentanyl for pain control
- MIDAZOLAM/FENTANYL: Midazolam for sedation and fentanyl for pain will be used for pleuroscopy monitored anesthesia care

SUMMARY:
The primary objective of this prospective trial will be to assess the effects of dexmedetomidine administration on oxygenation and respiratory function in patients undergoing diagnostic or therapeutic medical thoracoscopy/pleuroscopy for a pleural effusion compared to conventional conscious sedation/monitored anesthesia care (MAC) with midazolam. The secondary endpoint of the study will be to also assess the effects of dexmedetomidine administration on respiratory mechanics and postprocedural complications

DETAILED DESCRIPTION:
The study will be conducted at the Department of Anesthesiology and Pain Management in collaboration with the Department of Thoracic Surgery at the Attikon University Hospital, Athens.

The trial has received approval by the Attikon University Hospital's Scientific & Bioethics Committee and written informed consent will be obtained from all patients enrolled in the study.

Sample Size Calculation: A total of 60 patients will be assigned on a 1 to 1 basis to avoid bias to either a "DEX = dexmedetomidine" (n=30) or a "MIDAZOLAM/FENTANYL" group (n=30). To determine the required sample sizes quoted above, the statistical G-power calculator developed by Faul, Erdfelder, Lang, and Buchner was used. Values used to calculate the effect size (e=0.9326031) are based on results previously reported in the literature. For a study power of 90% with an alpha value of 0.05, a total of 26 patients in each group will need to be enrolled. Factoring in possible losses this number was rounded up to 30 patients per group.

Main Measurements Performance & Methods: Patients will initially be assessed with spirometry and arterial blood gas (ABG) analysis prior to the medical thoracoscopy/pleuroscopy to determine their baseline values of Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC) and Partial arterial Pressure of Oxygen/ Fraction of Inspiratory Oxygen (PaO2/FiO2) ratio respectively. Intra-operatively repeat ABG analysis will be performed at 30 minutes following the start of administration of the study drug. Subsequent to their medical thoracoscopy/pleuroscopy procedure study subjects will remain in the Post Anesthesia Care Unit (PACU) for a minimum of 1 hour following the discontinuation of the study drug. Repeated ABG analysis and spirometry will be carried out at that 1 hour to assess improvement over the pre-operative values. The administration of the spirometry exam will be by the same pulmonologist using the same spirometer device so as to minimize inter-observer variability. Arterial blood gas measurements will also be performed in the same analysis device.

Protocol for Sedation & Analgesia: Dexmedetomidine (DEX) group: Initial loading dose of dexmedetomidine will be 1.0 μg/kg of dexmedetomidine administered over 10 minutes. Fifteen minutes after starting the study drug administration, patients will be assessed for their level of sedation using the Observer's Assessment of Alertness/Sedation Scale (OAA/S), and any patient having a score ≥3 will receive intravenous (IV) midazolam in 0.5 mg doses, which will be repeated until the OAA/S is ≤2. MIDAZOLAM/FENTANYL group: Patients will be assessed for their level of sedation using the Observer's Assessment of Alertness/Sedation Scale (OAA/S), and any patient having a score ≥3 will receive intravenous (IV) midazolam in 0.5 mg doses, which will be repeated until the OAA/S is ≤2 All subjects will receive local anesthesia prior to the commencement of the "open" trocar insertion technique performed by the thoracic surgeon at the point of introduction of the rigid trocar in the pleural cavity with a combination of lidocaine 1.5% and ropivacaine 0.75%. If a patient is not adequately sedated, rescue midazolam will be administered as single IV boluses of 0.5 mg, which will be repeated as needed to achieve an OAA/S score of ≤3. Intravenous fentanyl, 25 μg boluses which can be repeated as necessary, will be given if a patient expresses a pain score of ≥3 during the study drugs infusion and ≥4 in the PACU on a Verbal scale of 0-10 (0 = no pain, 10 = worst pain), or if the anesthetist determines the presence of pain when verbal communication is not possible. Blood gas analysis will be obtained at 30' and 60' minutes intraoperatively. The dexmedetomidine infusion will be discontinued after wound closure.

At any time, if clinically indicated, the patient will be converted to an alternative sedative or anesthetic therapy and the study will be discontinued. OAA/S scores and all standard vital signs will be obtained every 5 min throughout the study drug infusion and before the administration of any rescue midazolam.

The time to reach OAA/S =5 from the end of infusion will be recorded. Other data recorded at the end of surgery will include total fentanyl and midazolam used intraoperatively, crystalloid infusion in litres, total mcg of the study drug (provided a [dex] = 4 mcg/ml) and postoperative Visual Analogue Scale (VAS) pain score. If VAS>3 acetaminophen 1 g will be administered. The patient's monitoring will be continued in the post-anesthesia care unit (PACU) with vital signs been recorded every 5 minutes for the first 15 minutes, then every 15 minutes for the next 45 minutes. Blood gas analysis will be obtained every 30' until discharge from the PACU. At 24 hours from the end of surgery, a spirometry will be performed. Patient satisfaction and surgeon satisfaction score will also be registered (4-point scale - 0 min to 3 max). Patients will be discharged from the PACU when their OAA/S score =5.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* American Society of Anesthesiologists (ASA) physical status of I-IV
* scheduled to undergo medical thoracoscopy/pleuroscopy.

Exclusion Criteria:

* general anesthesia within 7 days prior to study entry
* received an α2-agonist or antagonist within 14 days before the procedure
* received an intravenous opioid within 1 hour
* received an oral or intramuscular opioid within 4 hours from procedure
* New York Heart Association class ≥3
* acute unstable angina
* acute myocardial infarction (confirmed by laboratory findings) in the past 6 weeks
* heart rate (HR) ≤45-50 bpm
* systolic blood pressure (SBP) ≤90 mm Hg,
* 2nd or/and 3rd-degree Atrioventricular (AV) block (if the patient does not have a pacemaker)
* severe functional liver or kidney disease,
* obesity (body mass index ≥30 kg/m-2)
* severe restrictive interstitial lung disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who are scheduled for a pleuroscopy procedure.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
PaO2/FIO2 ratio | measured before procedure, every 30 minutes during procedure, before discharge from the postanesthesia care unit (approximately 2 hours after end of procedure)
  changes in lung oxygenation

SECONDARY OUTCOMES:
FEV1 (forced expiratory volume in 1 second) | before procedure and 24 hours after procedure
  respiratory mechanics
FVC (forced vital capacity) | before procedure and 24 hours after procedure
  respiratory mechanics
FEV1/FVC ratio | before procedure and 24 hours after procedure
  respiratory mechanics
PaCO2 | measured before procedure, every 30 minutes during procedure, before discharge from the postanesthesia care unit (approximately 2 hours after end of procedure)
  acid-base balance

OTHER OUTCOMES:
cumulative midazolam consumption | at the end of procedure
  measured in mg
cumulative fentanyl consumption | at the end of procedure
  measured in mg
cumulative dexmedetomidine consumption | at the end of procedure
  measured in mg
Observer's Assessment of Alertness/Sedation scale (OAA/S) | during procedure
  This 5 point Scale is used to assess level of sedation during the procedure (5- Responds readily to name spoken in normal tone, 4-Lethargic response to name spoken in normal tone, 3-Responds only after name is called loudly and/or repeatedly, 2-Responds only after mild prodding or shaking, 1-Does not respond to mild prodding or shaking)
Bradycardia | during the procedure
  incidence of bradycardia (HR <45 beats/ min) during procedure
Hypotension | during the procedure
  incidence of hypotension (MAP<65 mmHg) during procedure
Hypoxemia | during the procedure
  incidence of hypoxemia (SaO2< 92%) during procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Att, Athens, Greece